CLINICAL TRIAL: NCT00917813
Title: A Study of the Safety, Tolerability, and Pharmacokinetics of KD-247, a Humanized Monoclonal Antibody That Recognizes the Principal Neutralizing Determinant of HIV-1, in Asymptomatic HIV-1 Seropositive Individuals Who Are Not Receiving Concurrent Antiretroviral Therapy
Brief Title: A Study of Anti-HIV Monoclonal Antibody KD-247
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Chemo-Sero-Therapeutic Research Institute (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KD-1002
Record Dates: First submitted 2009-06-08; First posted 2009-06-10 (Estimated); Last update posted 2012-11-19 (Estimated); Status verified 2012-11

CONDITIONS: HIV Infections
Keywords: HIV; monoclonal antibody; KD-247; treatment naive
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- KD-247 (Experimental)
  Interventions: Drug: KD-247
- Placebo (Placebo Comparator)
  Interventions: Drug: Physiological saline

INTERVENTIONS:
Drug: KD-247 — Cohort 1 - 4 mg/kg KD-247 IV on Days 1, 8, and 15; Cohort 2 - 8 mg/kg KD-247 IV on Days 1, 8, and 15; Cohort 3 - 16 mg/kg KD-247 IV on Days 1, 8, and 15
  Arms: KD-247
Drug: Physiological saline — Cohort 1 - Physiological saline IV on Days 1, 8, and 15; Cohort 2 - Physiological saline IV on Days 1, 8, and 15; Cohort 3 - Physiological saline IV on Days 1, 8, and 15
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of 3 infusions of KD-247 over 2 weeks in HIV-1 seropositive individuals; to determine the pharmacokinetic parameters of KD-247 when administered as above; and to assess the effect of KD-247 infusions on plasma HIV-1 ribonucleic acid (RNA) load and on CD4+ T cell counts.

DETAILED DESCRIPTION:
A minimum of 6 active subjects and 3 placebo subjects for each dose cohort will complete 2 weeks of infusions. A maximum of 27 total subjects will be dosed with KD-247 and up to 9 total will receive placebo. Per cohort subjects randomized to active treatment will receive iv infusions of KD 247 over 2 hours at each dosing visit. Subjects randomized to placebo will receive 2-hour iv infusions of saline solution at each dosing visit. Following the first infusion of KD-247 (or placebo) for each subject in the study, there will be a 24-hour in-patient observation period before the next subject can be randomized within the study. Dose escalation will proceed only after safety data through Day 18 for all subjects in the lower-dose cohort is reviewed.

ELIGIBILITY:
Inclusion Criteria:

1. Have HIV-1 infection confirmed by enzyme immunoassay (EIA) and immunoblot.
2. Are male or female subjects, age 18-64 years.
3. Demonstrate an HIV-1 RNA copy number between 1000 and 100,000 copies/mL on 2 measurements at least 2 weeks apart. Measurements taken during screening and/or on a prior non-study related medical visit within 3 to 6 weeks of Study Day 1 may be considered.
4. Have CD4+ T cell count >350 cells/mm3 on 2 measurements at least 2 weeks apart. Measurements taken during screening and on one prior non-study medical visit within 3 to 6 weeks of Study Day 1 may be considered.
5. Are treatment naïve or have been off antiretroviral drugs for at least 8 weeks prior to screening.
6. By genotyping, have a sequence of the portion of the HIV envelope gene encoding the principal neutralizing determinant that is consistent with neutralization by KD-247.
7. Weigh 45-120 kg.
8. Have an absolute neutrophil count >1000 cells/uL, hemoglobin (Hgb) >10 g/dL, and platelets >100,000/uL.
9. Have serum creatinine ≤1.5 mg/dL and alanine transaminase (ALT) <2.5 times the upper limit of normal.
10. Have a 12-lead electrocardiogram (ECG) without clinically significant abnormalities in the opinion of the investigator.
11. Female subjects must be:

    * Women of non-childbearing potential, defined as either surgically sterile or at least 1-year post-menopausal (no menstrual periods for at least 2 years), or
    * Women of childbearing potential using a highly effective method of contraception, and
    * Women of childbearing potential with a negative serum beta human chorionic gonadotropin (β-HCG) test result at screening and within the 24 hours prior to administration of study drug. A negative urine pregnancy test within the 24 hours prior to administration of study drug will be acceptable, if the serum pregnancy test result is not yet available.
12. For heterosexual male subjects, the subject and the subject's sexual partner must agree to use acceptable methods of contraception during the entire study. Acceptable methods include, but are not limited to, intrauterine device, diaphragm with spermicide, condoms, or abstinence. Oral contraceptives alone are not an acceptable method of birth control.
13. Be willing and able to provide written informed consent.

Exclusion Criteria:

1. Have a history of an acquired immune deficiency syndrome (AIDS)-defining illness or symptomatic HIV disease (i.e., Centers for Disease Control [CDC] Class B or C).
2. Have received monoclonal antibody therapy of any kind in the past.
3. Received vaccinations in the past 15 days prior to study entry.
4. Received antihistamines in the 6 weeks prior to study entry.
5. Received non-steroidal anti-inflammatory drugs (NSAIDs) in the 5-6 days prior to skin test.
6. Any history of anaphylaxis, asthma, hypersensitivity reaction to a vaccine or drug infusion, angioedema, or urticaria.
7. Have been treated with any of the following within the 3 months prior to screening: interferons, cytokines, or other immunomodulators; immunoglobulin therapy; systemic corticosteroids; cytotoxic drugs; or ionizing radiation.
8. Have received any investigational agent within 60 days prior to screening.
9. Have any condition which, in the judgment of the investigator, may make the subject's participation in this study too risky; interfere with the collection of or interpretation of PK data; or interfere with the ability of the subject to adhere to and complete the study. Such conditions may include, but are not limited to, cardiovascular, respiratory, gastrointestinal/hepatic, neurologic, and genitourinary disorders.
10. Current alcohol or drug use that, in the judgment of the investigator, will interfere with the subject's ability to comply with the protocol requirements.
11. Have an unexplained positive urine drug screen test for an illicit drug.
12. Have a confirmed positive hepatitis B surface antigen (HBsAg) or antibody to hepatitis C virus (HCV).
13. Have used any prescription within 14 days of study initiation or any over-the-counter (OTC) medication within 3 days of study initiation which, in the judgment of the investigator, would place the individual at risk or interfere with safety, tolerability, or PK data.
14. Have dosages/amounts of drugs that have changed, or are scheduled to use new drugs which, in the judgment of the investigator, would place the individual at risk or interfere with safety, tolerability, or PK data.
15. Have a recent history of major surgery, internal organ biopsy, or major trauma.
16. Females who are pregnant or breast-feeding, or who plan to become pregnant during the study.
17. Have a mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study.
18. Show a positive reaction to the prick test for KD-247, i.e., ≥3 mm in diameter greater than the negative control.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Estimated)
Dates: Start 2007-09

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Pacific Oaks Medical Group, Beverly Hills, California
  - Providence Clinical Research, Burbank, California
  - Peter J. Ruane, MD, Inc., Los Angeles, California
  - Washington Hospital Center CAR, Washington D.C., District of Columbia
  - Gary Richmond, MD, PA, Fort Lauderdale, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Vita Research Solutions, Inc., Tamarac, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Northstar Medical, Chicago, Illinois
  - Institute of Human Virology, University of Maryland, Baltimore, Maryland
  - Albany Medical Center, Albany, New York
  - Aaron Diamond AIDS Research Center (ADARC), New York, New York
  - Central Texas Clinical Research, Austin, Texas
  - Therapeutic Concepts, P.A., Houston, Texas
  - DCOL Center for Clinical Research, Longview, Texas